CLINICAL TRIAL: NCT01068860
Title: A Multi-center, Double-blind, Placebo-controlled, Randomized Study to Compare the Effect of a Subcutaneous Canakinumab Administration to Placebo in Patients With Impaired Glucose Tolerance or Patients With Type 2 Diabetes Treated With Differing Baseline Diabetes Therapies
Brief Title: To Compare the Effect of a Subcutaneous Canakinumab Administration to Placebo in Patients With Impaired Glucose Tolerance or Patients With Type 2 Diabetes With Differing Baseline Diabetes Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885I2207
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes Mellitus; Impaired Glucose Tolerance
Keywords: Type 2 Diabetes Mellitus; canakinumab; Pre diabetic; glucose intolerant; oral anti diabetic medication; insulin treatment; metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Metabolic Syndrome | interventions — canakinumab; Metformin; Chlorpropamide; Acetohexamide; Tolazamide; Tolbutamide; Glipizide; glimepiride; Glyburide; Troglitazone; Insulin; Insulin, Regular, Pork; Insulin Lispro; Insulin, Regular, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Canakinumab 150 mg + Metformin (Experimental): Eligible participants received a single subcutaneous injection Canakinumab 150 mg.Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) monotherapy treatment at least 1000 mg/day for 3 months prior to screening
  Interventions: Drug: Canakinumab 150 mg
- Placebo + Metformin (Placebo Comparator): Eligible participants received a single subcutaneous injection of Placebo to Canakinumab. Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) monotherapy treatment at least 1000 mg/day for 3 months prior to screening
  Interventions: Drug: Placebo to Canakinumab
- Canakinumab 150 mg + Metforimin + Sulfonylurea (Experimental): Eligible participants received a single subcutaneous injection of Canakinumab 150 mg.Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) at least 1000 mg/day , and a Sulfonylurea (Sulfonyl), at least 1/2 the maximally labeled dose combination therapy, for 3 months prior to screening.
  Interventions: Drug: Canakinumab 150 mg
- Placebo + Metforimin + Sulfonylurea (Placebo Comparator): Eligible participants received a single subcutaneous injection of Placebo to Canakinumab.Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) at least 1000 mg/day , and a Sulfonylurea (Sulfonyl), at least 1/2 the maximally labeled dose combination therapy, for 3 months prior to screening.
  Interventions: Drug: Placebo to Canakinumab
- Canakinumab 150 mg + Met + Sulfonyl + Thiazolidinedione (Experimental): Eligible participants received a single subcutaneous injection of Canakinumab 150 mg.Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) at least 1000 mg/day , and a Sulfonylurea (Sulfonyl), at least 1/2 the maximally labeled dose, and a Thiazolidinedione (Thiaz)at least 1/2 the maximally labeled dose combination therapy, for 3 months prior to screening.
  Interventions: Drug: Canakinumab 150 mg
- Placebo + Met + Sulfonyl + Thiazolidinedione (Placebo Comparator): Eligible participants received a single subcutaneous injection of Placebo to Canakinumab. Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) at least 1000 mg/day , and a Sulfonylurea (Sulfonyl), at least 1/2 the maximally labeled dose, and a Thiazolidinedione (Thiaz)at least 1/2 the maximally labeled dose combination therapy, for 3 months prior to screening.
  Interventions: Drug: Placebo to Canakinumab
- Canakinumab 150 mg + Insulin (Experimental): Eligible participants received a single subcutaneous injection of Canakinumab 150 mg. Patients must have had documented diagnosis of Type 2 Diabetes Mellitus for 3 months prior to screening and be on a stable dose of Insulin, 2 insulin injections per day for a total daily dose of less than 100 U with or without Metformin (Met)for 3 months prior to screening
  Interventions: Drug: Canakinumab 150 mg
- Placebo + Insulin (Placebo Comparator): Eligible participants received a single subcutaneous injection of Placebo to Canakinumab. Patients must have had documented diagnosis of Type 2 Diabetes Mellitus for 3 months prior to screening and be on a stable dose of Insulin, 2 insulin injections per day for a total daily dose of less than 100 U with or without Metformin (Met)for 3 months prior to screening
  Interventions: Drug: Placebo to Canakinumab
- Canakinumab 150 mg in patients with IGT (Experimental): Eligible participants received a single subcutaneous injection of Canakinumab 150 mg. Patients must have had Impaired Glucose Tolerance (IGT) as defined by the World Health Organization (WHO) criteria confirmed at screening visit.
  Interventions: Drug: Canakinumab 150 mg
- Placebo in patients with IGT (Placebo Comparator): Eligible participants received a single subcutaneous injection of Placebo to Canakinumab. Patients must have had Impaired Glucose Tolerance (IGT) as defined by the World Health Organization (WHO) criteria confirmed at screening visit.
  Interventions: Drug: Placebo to Canakinumab

INTERVENTIONS:
Drug: Canakinumab 150 mg — Single subcutaneous injection of Canakinumab 150 mg.
  Other Names: ACZ885; Glucophage; Chlorpropramide; Diabinese; Acetohexamide; Dymelor; Tolazamise; Tolinase; Tolbutamise; Orinase; Glipizide; Glucotrol; Glimepiride; Amaryl; Glyburide; DiaBeta; Micronase; Glynase PresTab; Troglitazone; Rezulin; Insulin; Iletin; Novolin; Velosulin; Humalog; Humulin; Lente; Ultralente; NPH Iletin
  Arms: Canakinumab 150 mg + Insulin; Canakinumab 150 mg + Met + Sulfonyl + Thiazolidinedione; Canakinumab 150 mg + Metforimin + Sulfonylurea; Canakinumab 150 mg + Metformin; Canakinumab 150 mg in patients with IGT
Drug: Placebo to Canakinumab — Single subcutaneous injection of Placebo to Canakinumab.
  Other Names: ACZ885; Glucophage; Chlorpropramide; Diabinese; Acetohexamide; Dymelor; Tolazamise; Tolinase; Tolbutamise; Orinase; Glipizide; Glucotrol; Glimepiride; Amaryl; Glyburide; DiaBeta; Micronase; Glynase PresTab; Troglitazone; Rezulin; Insulin; Iletin; Novolin; Velosulin; Humalog; Humulin; Lente; Ultralente; NPH Iletin
  Arms: Placebo + Insulin; Placebo + Met + Sulfonyl + Thiazolidinedione; Placebo + Metforimin + Sulfonylurea; Placebo + Metformin; Placebo in patients with IGT

SUMMARY:
This was a 10-week, placebo-controlled, randomized study to investigate the effect of injectable IL-1B antagonist, Canakinumab , in participants with impaired glucose tolerance or Type 2 Diabetes Mellitus (T2DM) already treated on different background diabetes therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must fulfill all criteria in one of the following groups:

   * Impaired Glucose Tolerance (IGT) as diagnosed per protocol and not on an anti-diabetic medicine during the study
   * Diagnosis of Type 2 diabetes in stable treatment with metformin
   * Diagnosis of Type 2 diabetes in stable treatment with metformin (at least 1000 mg/day) in combination with a sulfonylurea
   * Diagnosis of Type 2 diabetes in stable treatment with metformin (at least 1000 mg/day), sulfonylurea and thiazolidinedione combination therapy
   * Diagnosis of Type 2 diabetes in stable treatment with at least two insulin injections a day with or without metformin
2. HbA1c between 6.5% and 8%, inclusive, at Screening; this criterion does not apply to the IGT group
3. Age from 18-74 years, inclusive, and of either sex

Exclusion Criteria:

1. Type 1 diabetes or diabetes that is a result of pancreatic injury or other secondary forms of diabetes
2. History or current findings of active pulmonary disease (e.g. tuberculosis, fungal diseases) as defined in the protocol:
3. Known presence or suspicion of active or recurrent bacterial, fungal or viral infection at the time of enrollment proven.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corporation, Study Director — Novartis Pharmaceuticals
Locations (52):
- United States (11):
  - National Research Institute, Los Angeles, California
  - Crest Clinical Trials, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Commonwealth Biomedical Research LLC, Madisonville, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - VA Medical Center, Omaha, Nebraska
  - Lillestol Research LLC, Fargo, North Dakota
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Texas Center for Drug Development P.A., Houston, Texas
  - Utah Clinical Trials, Salt Lake City, Utah
- Australia (3):
  - Barwon Health - Geelong Hospital, Geelong, Victoria
  - Austin Health - Heidelberg Repatriation Hospital, Heidelberg Heights, Victoria
  - Melbourne Health - Royal Melbourne Hospital, Melbourne, Victoria
- Canada (5):
  - Lifestyle Metabolism Centre (Etobicoke), Etobicoke, Ontario
  - LMC Endocrinology Centres (Markham) Ltd, Markham, Ontario
  - LMC Endocrinology Centres (Thornhill) Ltd, Thornhill, Ontario
  - Centre de recherche clinique de Laval, Laval, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
- Finland (3):
  - Lihavuustutkimusyksikkö, Helsinki
  - Lääkärikeskus Mehiläinen Töölö, Helsinki
  - ODL Terveys Oy, Oulu
- Germany (14):
  - Clintrial Berlin Praxis fuer medizinische Studien, Berlin
  - Klinische Forschung Berlin-Buch Dr. Andrei Khariouzov, Berlin
  - Gemeinschaftspraxis Dr. Ingo Zeissig, Duisburg
  - "Sana Krankenhaus Gerresheim, Düsseldorf
  - Praxis Dr. Thorsten Rau, Essen
  - Praxis Dr. med. Joerg Luedemann, Falkensee
  - Dr. Helmut Anderten Gemeinschaftspraxis Dres. Anderten und Krok, Hildesheim
  - Praxis Dr. Julia Chevts, Karlsruhe
  - Pro Scientia Med, Lübeck
  - Praxis Dr. Winfried Keuthage, Münster
  - Praxis Dr. Uwe Boeckmann, Neumünster
  - Dr. Klaus Funke IkFE Studiencenter Potsdam GMBH I.G., Potsdam
  - Praxis Dr. Gerhard Steinmaier, Viernheim
  - Praxis Dr. Reinhold U. Schneider, Wetzlar-Naunheim
- India (8):
  - Visakha Diabetes & Endocrine Centre, Visakhapatnam, Andhra Pradesh
  - Jnana Sanjeevini Medical Center, Bangalore, Kar
  - Bangalore Diabetes Hospital,, Banglore, KAR
  - Health & Research Centre, Trivandrum, Ker
  - Diabetes Thyroid Hormone Research Institute Pvt .Ltd., Indore, Madhya Pradesh
  - Indrayani Speciality Hospital,, Nagpur, Maharashtra
  - Sahyadri Hospital Bibewewadi Centre of Excellence for Diabetics, Pune, Mah
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
- Italy (8):
  - Azienda Ospedaliera-Ospedali Riuniti di BergamoU, Bergamo, BG
  - Az. Ospedaliera Universit. S.Martino-Universita degli Studi, Genova, GE
  - Azienda Ospedaliera S. Paolo-Polo Universitario, Milan, MI
  - Fondazione Centro San Raffaele del Monte Tabor-IRCCSUnità, Milan, Mi
  - Az. Ospedaliera Della Prov.di Pavia, Casorate Primo, PV
  - Policlinico A.Gemelli - Univ.Cattolica del Sacro Cuore, Roma, Roma
  - A.O.Universitaria Senese, Universita degli Studi di Siena, Siena, SI
  - S.C.D.U. Endocrinologia e Malattie del Metabolismo, Torino, To

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Qualified patients entered a 4-week run-in period while taking current therapy thru the study. After the run-in, patients had the baseline meal challenge. Then patients were randomized. A 2nd meal challenge was performed after 4 wks. This ended the study except for a follow up phone call after approx.90 days to record serious adverse events (SAEs)
Groups:
- Canakinumab 150 mg + Metformin: Eligible participants received a single subcutaneous injection Canakinumab 150 mg. Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) monotherapy treatment at least 1000 mg/day for 3 months prior to screening
- Canakinumab 150 mg + Metformin + Sulfonylurea: Eligible participants received a single subcutaneous injection of Canakinumab 150 mg.Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) at least 1000 mg/day , and a Sulfonylurea (Sulfonyl), at least 1/2 the maximally labeled dose combination therapy, for 3 months prior to screening.
- Placebo + Metformin + Sulfonylurea: Eligible participants received a single subcutaneous injection of Placebo to Canakinumab.Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) at least 1000 mg/day , and a Sulfonylurea (Sulfonyl), at least 1/2 the maximally labeled dose combination therapy, for 3 months prior to screening.
- Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia: Eligible participants received a single subcutaneous injection of Canakinumab 150 mg.Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) at least 1000 mg/day , and a Sulfonylurea (Sulfonyl), at least 1/2 the maximally labeled dose, and a Thiazolidinedione (Thiaz)at least 1/2 the maximally labeled dose combination therapy, for 3 months prior to screening.
- Placebo + Met + Sulfonyl + Thiaz: Eligible participants received a single subcutaneous injection of Placebo to Canakinumab. Patients must have had documented diagnosis of Type 2 Diabetes Mellitus and be on a stable dose of Metformin (Met) at least 1000 mg/day , and a Sulfonylurea (Sulfonyl), at least 1/2 the maximally labeled dose, and a Thiazolidinedione (Thiaz)at least 1/2 the maximally labeled dose combination therapy, for 3 months prior to screening.
- Canakinumab 150 mg in Participants With IGT: Eligible participants received a single subcutaneous injection of Canakinumab 150 mg. Patients must have had Impaired Glucose Tolerance (IGT) as defined by the World Health Organization (WHO) criteria confirmed at screening visit.
- Placebo in Participants With IGT: Eligible participants received a single subcutaneous injection of Placebo to Canakinumab. Patients must have had Impaired Glucose Tolerance (IGT) as defined by the World Health Organization (WHO) criteria confirmed at screening visit.
Period: Overall Study
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Started | 33 | 17 | 33 | 17 | 32 | 16 | 28 | 15 | 28 | 27
Completed | 33 | 16 | 33 | 16 | 32 | 14 | 28 | 15 | 28 | 23
Not Completed | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3
Not completed — Administrative problems; misrandomized | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT | Total
Number analyzed (Participants) | 33 | 17 | 33 | 17 | 32 | 16 | 28 | 15 | 28 | 27 | 246
Age, Customized [Mean (Standard Deviation); unit: years] | 55.9 (10.50) | 56.5 (9.30) | 60.0 (8.17) | 59.4 (8.02) | 59.1 (10.63) | 57.2 (9.39) | 58.6 (10.11) | 57.0 (13.86) | 52.8 (10.90) | 57.6 (10.07) | 57.4 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 3 | 14 | 10 | 11 | 5 | 13 | 10 | 12 | 16 | 113
  Male | 14 | 14 | 19 | 7 | 21 | 11 | 15 | 5 | 16 | 11 | 133

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Meal Stimulated Insulin Secretion Rate (ISR) Relative to Glucose 0-2 Hours, From Baseline to 4 Weeks.
Description: Change in Insulin Secretion Rate stimulated by Liquid mixed-meal challenge. Blood samples were taken prior to and after meal for glucose and insulin at sample times: -20, -10, -1 and 10, 20, 30, 60, 90, 120, 180, and 240 minutes relative to the start of the meal.A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include patients from the IGT population
Time Frame: Baseline, 4 weeks
Population: Participants from the full analysis set who participated in the meal challenge and who had at least 1 post-baseline absolute glucose measurement at 2 hours.
Measure: Least Squares Mean (Standard Error); unit: pmol/min/m^2/mmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 16 | 31 | 15 | 31 | 14 | 26 | 15 | 28 | 21
pmol/min/m^2/mmol/L | -0.06 (0.943) | -0.23 (1.334) | 0.04 (0.958) | 0.45 (1.378) | -0.79 (0.958) | 1.16 (1.426) | 1.23 (1.046) | -0.49 (1.378) | -1.50 (1.975) | -1.93 (1.737)

2. Secondary Outcome: Mean Change in Meal Stimulated Insulin Secretion Rate (ISR) Relative to Glucose 2-4 Hours, From Baseline to 4 Weeks
Description: Change in Insulin Secretion Rate stimulated by Liquid mixed-meal challenge Blood samples were taken prior to and after meal for glucose and insulin at sample times: -20, -10, -1 and 10, 20, 30, 60, 90, 120, 180, and 240 minutes relative to the start of the meal. A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/min/m^2/mmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 16 | 30 | 15 | 31 | 14 | 26 | 15 | 28 | 20
pmol/min/m^2/mmol/L | 0.21 (2.000) | -2.15 (2.829) | -2.98 (2.066) | 2.02 (2.921) | 0.15 (2.032) | 1.19 (3.024) | -0.43 (2.219) | -0.51 (2.921) | -0.71 (1.040) | -1.00 (1.518)

3. Secondary Outcome: Mean Change in Meal Stimulated Insulin Secretion Rate (ISR) Relative to Glucose 0-4 Hours, From Baseline to 4 Weeks.
Description: Change in Insulin Secretion Rate stimulated by Liquid mixed-meal challenge. Blood samples were taken prior to and after meal for glucose, insulin and C-peptide at sample times: -20, -10, -1 and 10, 20, 30, 60, 90, 120, 180, and 240 minutes relative to the start of the meal. A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/min/m^2/mmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 33 | 16 | 31 | 15 | 32 | 14 | 26 | 15 | 28 | 21
pmol/min/m^2/mmol/L | 0.44 (0.858) | -0.99 (1.232) | -0.32 (0.885) | 1.22 (1.272) | -0.63 (0.871) | 1.24 (1.317) | 0.53 (0.966) | -0.49 (1.272) | -1.38 (1.356) | -1.35 (1.330)

4. Secondary Outcome: Mean Change in Fasting Plasma Glucose, From Baseline to 4 Weeks
Description: Change in Fasting Glucose Level measured from plasma taken at Baseline and after 4 weeks of treatment.
  A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 33 | 16 | 31 | 16 | 32 | 14 | 26 | 15 | 28 | 21
mmol/L | -0.32 (0.272) | 0.33 (0.391) | -0.20 (0.281) | -0.23 (0.391) | -0.33 (0.276) | -0.36 (0.418) | -0.26 (0.307) | -0.80 (0.404) | -0.06 (0.107) | 0.10 (0.094)

5. Secondary Outcome: Mean Change in Fructosamine, From Baseline to 4 Weeks
Description: Change in Fructosamine Level taken from plasma, measured at Baseline and after 4 weeks of treatment.
  A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 33 | 16 | 31 | 16 | 32 | 14 | 27 | 15 | 28 | 23
mmol/L | -5.30 (3.727) | -0.75 (5.353) | -3.45 (3.846) | -7.50 (5.353) | -1.81 (3.785) | -3.07 (5.722) | -3.00 (4.121) | -19.73 (5.528) | -6.36 (3.259) | 1.39 (3813)

6. Secondary Outcome: Mean Change in Fasting Plasma Insulin, From Baseline to 4 Weeks
Description: Change in Fasting Insulin level taken from plasma, measured at Baseline and after 4 weeks of treatment.
  A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 33 | 15 | 30 | 15 | 31 | 13 | 26 | 15 | 28 | 23
pmol/L | -3.58 (8.703) | 10.73 (12.908) | -16.07 (9.128) | -9.40 (12.908) | -0.77 (8.979) | 2.31 (13.866) | 21.27 (9.805) | 25.67 (12.908) | -.021 (6.093) | -3.43 (4.554)

7. Secondary Outcome: Mean Change in Quantitative Insulin Sensitivity Check Index (QUICKI) Score, From Baseline to 4 Weeks
Description: The Quantitative Insulin Sensitivity Check Index (QUICKI) score, measures insulin sensitivity which is the inverse of insulin resistance. The score is calculated by the equation: 1 /(log(fasting insulin µU/mL) + log(fasting glucose mg/dL)). In normal subjects the mean score ± SE is 0.366 ± 0.029.
  A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: number
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 33 | 15 | 30 | 15 | 31 | 13 | 25 | 15 | 28 | 21
number | 0.004 (0.0080) | -0.000 (0.0119) | 0.002 (0.0084) | 0.009 (0.0119) | 0.018 (0.0083) | -0.001 (0.0128) | -0.003 (0.0092) | 0.005 (0.0119) | -0.001 (0.0051) | 0.001 (0.0034)

8. Secondary Outcome: Mean Change in Fasting Glucose Disposition Index(GDI)1 and Index 2, From Baseline to 4 Weeks
Description: GDI 1 is the product of insulin sensitivity index (Si)during the 1st phase of insulin secretion and β-cell function as measured by the acute insulin response (AIR).GDI 2 is the product of (Si)during the 2nd phase of insulin secretion and β-cell function as measured by the acute insulin response (AIR). A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT group.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: number
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 15 | 30 | 15 | 30 | 13 | 25 | 15 | 26 | 21
number
  Index 1 | 0.06 (0.374) | -0.29 (0.546) | 0.06 (0.386) | 0.37 (0.546) | 0.24 (0.386) | 0.33 (0.586) | 0.25 (0.423) | -0.27 (0.546) | -0.51 (0.672) | -0.64 (0.530)
  Index 2 (n= 32,15, 29,15, 30,13, 25, 15, 20, 26) | 0.14 (0.652) | -0.81 (0.952) | -0.94 (0.685) | 0.81 (0.952) | 0.62 (0.673) | 0.49 (1.023) | -0.21 (0.738) | -0.25 (0.952) | -0.16 (0.396) | -0.31 (0.509)

9. Secondary Outcome: Mean Change in Absolute Glucose Level at 2 Hours, From Baseline to 4 Weeks
Description: Change in glucose level measured after 2 hours of fasting. Blood sample was drawn at 0 minutes and at 240 minutes.
  A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 16 | 31 | 15 | 31 | 14 | 26 | 15 | 28 | 21
mmol/L | -0.53 (0.389) | 0.13 (0.551) | -0.60 (0.396) | 0.18 (0.551) | -1.08 (0.396) | -0.56 (0.589) | -0.56 (0.432) | -0.16 (0.569) | -0.26 (0.241) | -0.25 (0.213)

10. Secondary Outcome: Mean Change in Insulin Area Under the Curve (AUC) 0-4 Hours, From Baseline to 4 Weeks
Description: Blood samples were drawn after a test meal at 0, 15, 30, 45, 60, 90, 120, 180 and 240 min. Insulin levels over 4 hrs were shown as Area Under the Curve,(AUC). AUC was calculated as: x=1 AUC ΣAx n Where Ax = AUC for the 240 min.interval, and X = 1 for the 1st interval. A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab vs placebo within each T2DM group. The mixed model didn't include the IGT group.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol*hour/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 16 | 31 | 15 | 31 | 14 | 26 | 15 | 28 | 21
pmol*hour/L | -9.37 (40.538) | 1.21 (60.128) | -73.25 (42.517) | -38.32 (60.128) | -36.96 (41.825) | 8.46 (64.587) | 163.87 (45.670) | 139.24 (60.128) | 44.27 (60.700) | -106.68 (53.615)

11. Secondary Outcome: Mean Change in C-peptide Area Under the Curve (AUC), 0-4 Hours, From Baseline to 4 Weeks
Description: as for outcome 10
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol*hour/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 16 | 31 | 15 | 31 | 14 | 26 | 15 | 28 | 21
nmol*hour/L | -0.18 (0.225) | -0.18 (0.324) | -0.21 (0.232) | 0.12 (0.334) | -0.61 (0.229) | 0.02 (0.346) | 0.16 (0.249) | -0.29 (0.334) | -0.43 (0.253) | -0.40 (0.288)

12. Secondary Outcome: Mean Change in Post-prandial Glucose Area Under the Curve (AUC)0-4 Hours, From Baseline to 4 Weeks
Description: as for outcome 10
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol*hr/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 16 | 31 | 15 | 31 | 14 | 26 | 15 | 28 | 21
mmol*hr/L | -0.59 (1.296) | 0.46 (1.861) | -1.37 (1.337) | -1.24 (1.861) | -3.58 (1.316) | -2.88 (1.990) | -1.49 (1.460) | -1.76 (1.922) | -0.71 (0.554) | -0.10 (0.512)

13. Secondary Outcome: Mean Change in Peak Plasma Glucose, From Baseline to 4 Weeks
Description: Change in peak plasma glucose level as measured from Baseline to 4 weeks of treatment.
  A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 16 | 31 | 15 | 31 | 14 | 26 | 15 | 28 | 21
mmol/L | -0.41 (0.369) | 0.21 (0.531) | -0.43 (0.381) | -0.03 (0.531) | -0.82 (0.375) | -0.77 (0.567) | -0.15 (0.416) | -0.60 (0.548) | -0.34 (0.181) | -0.04 (0.189)

14. Secondary Outcome: Mean Change in Peak Plasma Insulin, From Baseline to 4 Weeks
Description: Change in mean peak plasma Insulin level as measured from Baseline to 4 weeks of treatment. A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 16 | 31 | 15 | 31 | 14 | 26 | 15 | 28 | 21
pmol/L | 8.09 (22.673) | 44.56 (32.561) | -55.07 (23.779) | 11.33 (33.629) | 5.13 (23.392) | -5.15 (36.123) | 91.74 (25.065) | 36.87 (33.629) | 56.21 (27.952) | -26.43 (40.163)

15. Secondary Outcome: Mean Change in Peak Plasma C-peptide Level, From Baseline to 4 Weeks
Description: Change in mean peak plasma C-peptide level measured from Baseline to 4 weeks of treatment.
  A mixed model with treatment fitted as fixed effect, and population and the interaction of population and treatment fitted as random effects were used for the comparison of Canakinumab versus placebo within each T2DM population. The mixed model did not include participants from the IGT population.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 32 | 16 | 31 | 15 | 31 | 14 | 26 | 15 | 28 | 21
nmol/L | -0.04 (0.081) | -0.04 (0.116) | -0.10 (0.083) | 0.16 (0.120) | -0.21 (0.082) | 0.05 (0.124) | 0.07 (0.089) | -0.14 (0.120) | -0.18 (0.101) | -0.18 (0.134)

16. Secondary Outcome: Number of Participants Reporting Death, Serious Adverse Events (SAEs) and Adverse Events (AEs) Above 5% Frequency, From Baseline to 4 Weeks
Description: An adverse event is any unwanted event, whether related to study drug or not occuring during the study period. A Serious Adverse Event (SAE) is an event resulting in death, requiring or prolonging hospitalization, a congenital anomaly or other important medical event. AEs and SAEs were recorded at each visit.
Time Frame: Baseline, 4 weeks
Population: Safety Population consisted of all participants who received at least one dose of study medication and had at least one post-baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metformin + Sulfonylurea | Placebo + Metformin + Sulfonylurea | Canakinumab 150 mg Canakinumab 150 mg + Met + Sulfonyl + Thia | Placebo + Met + Sulfonyl + Thiaz | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Participants With IGT | Placebo in Participants With IGT
Number analyzed (Participants) | 33 | 17 | 32 | 17 | 32 | 16 | 28 | 15 | 28 | 26
participants
  Number of Participants with Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of Participants with Non-serious AEs > 5% | 0 | 4 | 6 | 3 | 4 | 3 | 6 | 3 | 0 | 0

ADVERSE EVENTS:
Description: Safety Set included all randomized participants who received study drug.
Arm/Group | Canakinumab 150 mg + Metformin | Placebo + Metformin | Canakinumab 150 mg + Metforimin + Sulfonylurea | Placebo + Metforimin + Sulfonylurea | Canakinumab 150 mg + Met + Sulfonyl + Thiazolidinedione | Placebo + Met + Sulfonyl + Thiazolidinedione | Canakinumab 150 mg + Insulin | Placebo + Insulin | Canakinumab 150 mg in Patients With IGT | Placebo in Patients With IGT
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/17 | 0/32 | 0/17 | 0/32 | 0/16 | 0/28 | 0/15 | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 0/33 | 4/17 | 6/32 | 3/17 | 4/32 | 3/16 | 6/28 | 3/15 | 0/28 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab 150 mg + Metformin (N=33) | Placebo + Metformin (N=17) | Canakinumab 150 mg + Metforimin + Sulfonylurea (N=32) | Placebo + Metforimin + Sulfonylurea (N=17) | Canakinumab 150 mg + Met + Sulfonyl + Thiazolidinedione (N=32) | Placebo + Met + Sulfonyl + Thiazolidinedione (N=16) | Canakinumab 150 mg + Insulin (N=28) | Placebo + Insulin (N=15) | Canakinumab 150 mg in Patients With IGT (N=28) | Placebo in Patients With IGT (N=26)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Antinuclear antibody positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.